CLINICAL TRIAL: NCT01529489
Title: Effect of the Combined (Aerobic/Resisted) and Interval Physical Training on Oxygen Uptake and Heart Rate On-kinetics Responses in Patients With Moderate to Very Severe COPD: Double-blind, Randomized, Controlled Trial
Brief Title: Effect of Two Physical Training Programs on Oxygen Uptake and Heart Rate On-kinetics in Patients COPD
Acronym: BVPS-123
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Sao Carlos (Other)
Responsible Party: Principal Investigator, Bruna Varanda Pessoa, Principal Investigator, Universidade Federal de Sao Carlos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BVPS-123
Record Dates: First submitted 2012-02-02; First posted 2012-02-08 (Estimated); Last update posted 2012-02-08 (Estimated); Status verified 2012-02

CONDITIONS: Chronic Obstructive Pulmonary Disease; Healthy
Keywords: Chronic Obstructive Pulmonary Disease; Physical training; Oxygen uptake kinetic; Heart rate kinetic
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Interval physical training Control group (Active Comparator)
  Interventions: Other: Interval physical training in elliptical equipament
- Resisted/Aerobic physical training group (Experimental)
  Interventions: Other: Resisted/Aerobic physical training
- Aerobic/resisted physical training group (Active Comparator)
  Interventions: Other: Resisted/Aerobic physical training
- Interval physical training group (Experimental): COPD, interval physical training, elliptical equipament, oxygen uptake kinetic, heart rate kinetic
  Interventions: Other: Interval physical training in elliptical equipament

INTERVENTIONS:
Other: Resisted/Aerobic physical training — COPD, aerobic physical training in cicloergometer, resisted physical training in cicloergometer, oxygen uptake kinetic, heart rate kinetic.
  Other Names: COPD,; aerobic physical training in cicloergometer,; resisted physical training in cicloergometer,; oxygen uptake kinetic,; heart rate kinetic.
  Arms: Resisted/Aerobic physical training group
Other: Interval physical training in elliptical equipament — Control group (healthy individuals), interval physical training, elliptical equipment, oxygen uptake kinetic, heart rate kinetic.
  Other Names: Control group (healthy individuals),; interval physical training in elliptical equipment,; oxygen uptake kinetic,; heart rate kinetic.
  Arms: Interval physical training Control group
Other: Interval physical training in elliptical equipament — COPD, interval physical training, elliptical equipament, oxygen uptake kinetic, heart rate kinetic
  Other Names: COPD,; interval physical training in elliptical equipament,; oxygen uptake kinetic,; heart rate kinetic.
  Arms: Interval physical training group
Other: Resisted/Aerobic physical training — Control group, aerobic physical training in cicloergometer, resisted physical training in leg-press oxygen uptake kinetic heart rate kinetic
  Other Names: Control group,; aerobic physical training in cicloergometer,; resisted physical training in leg-press,; oxygen uptake kinetic,; heart rate kinetic.
  Arms: Aerobic/resisted physical training group

SUMMARY:
Patients with chronic obstructive pulmonary disease (COPD) present slowed pulmonary oxygen uptake (VO2) and heart rate (HR) kinetics compared with age-matched controls. Patients with COPD present significant loss of body mass, decreased strength and endurance of respiratory muscles and lower limbs, leading reduced exercise capacity. This reduced exercise capacity can be marked by slowed kinetics of VO2 and HR at the onset of heavy-intensity exercise. Additionally, derangements in the diffusive and convective transport of oxygen to skeletal muscle mitocondria, and intramyocyte metabolic machinery, higher ventilation and disturbances in mechanics of breathing, hypoxemia, pulmonary hemodynamics, autonomic balance, and peripheral vasodilation, and accumulation of by-products that might be related to increased muscle fatigability could slow the response of systemic (central) and peripheral (microvascular) oxygen delivery to a point where the kinetics of VO2 might become limited by O2 availability and HR. Thus, the physical training programs of the lower limbs, in addition to presenting scientific evidence "A", are important components, resulting in the reversal of the manifestations of COPD, resulting in improvement in exercise capacity, well significantly speeded VO2 and HR kinetics in patients with COPD. However, it should be taken into account the choice of an appropriate program limitations and severity of disease. Assuming that COPD patients present slower VO2 and HR kinetics, the investigators hypothesized that the heavy-intense interval physical training in equipament elliptical would promote a greater increase in the functionality (functional performance) and speeded kinetics in the cycle ergometer and elliptical equipment constant-load intense exercises tests of COPD patients. In this context, the present study intends to evaluate and compare the effects of resistive plus aerobic physical training and interval physical training on oxygen consumption (VO2) and heart rate (HR) kinetics responses at the onset in cycle ergometer and elliptical equipment constant-load intense exercises tests in patients with COPD.

DETAILED DESCRIPTION:
Subjects performed after and before of two physical training program the following tests: lung function test,cardiopulmonary exercise testing (CPT), constant-load exercise test in cycle ergometer, Constant-load exercise test in elliptical equipament, one repetition maximum test(1RM), on alternate days.

* Lung function: All patients underwent spirometry with the determination of FEV1 and FVC according to American Thoracic Society recommendations. Spirometry was performed using a COSMED microQuark PC - based Spirometer ®, (Pavona di Albano - Roma, Itália), which was calibrated before each test.
* Cardiopulmonary Exercise Testing (CPT): Incremental symptom-limited exercise testing was performed on a cycle-ergometer(Ergo FIT®, model Ergo 167 Cycle, Pirmasens, Germany) using a computer-based ventilatory expired gas analysis system (VO2000, Medgraphics Corp., St. Paul, MN). All subjects underwent a CPT to determine the peak work rate and the peak oxygen uptake (peak VO2). The subjects' electrocardiographic recordings were monitored using a cardiac monitor, SpO2, BP and sensation of dyspnea and fatigue using the BE-CR-10. A gas analyzer (VO2000 Medgraphics®, St Paul MN, USA) was used to obtain the participants' VO2 at each stage of the test. The ergospirometric values were recorded by the mean value measured every three breaths using the Aerograph® program. The VO2 was determined choosing the higher and more coherent value in the final 30 seconds of each stage.
* Constant-load exercise test in cycle ergometer and Constant-load exercise test in elliptical equipament: The two exercise tests were performed at 70% of the previously determined work rate in CPT. During the CSET, VO2 was measured breath-by-breath and averaged every three respiration, while SpO2, HR, and the electrocardiogram were continuously monitored, and calculated a on-Kinetics of VO2 and HR.

  * Physical training program:
* The interval physical training on the elliptical trainer (Kiko's® HM 6022, São Paulo, SP, Brazil) totalized 18 sessions that the individuals of both groups had to attend at least twice a week. Each session lasted not more than 60 minutes and they were all individual meetings. The minimal work rate of the equipment was 40W and the lower increment work rate was 10W. The elliptical trainer allowed combined exercise with the upper limb, however, in the present study, the exercise was performed with the arms fixed, and every participant's HR was monitored using a pulse frequency meter (Polar® FS2cTM Kempele, Finland), the pulse oxygen saturation (SpO2) using a pulse oximeter (Nonin®, model 8500A, Minneapolis, Mn, USA), the blood pressure (BP) using a mercury sphygmomanometer (Oxigel®, São Paulo, SP, Brazil) and the sensation of dyspnea and lower limb fatigue using the Modified Borg CR-10 Scale (BE-CR10). The elliptical exercise was an interval training and was based on studies that performed interval training exercise in cycle ergometer. This was a 30-minute exercise with a rest interval established in one minute. The exercise's work rateworkload was the maximal achieved in the CPT, and it was not modified until the sessions were finished The individuals who did not reach 40W in the CPT performed 30 seconds exercising periods at 40W with 1-minute resting interval. The volunteers who achieved workload equal or higher 40W performed 1-minute exercising periods at the workload achieved in the CPT with 1-minute resting interval. During the exercise on the equipment, the individuals should keep the speed between 40 and 50 rpm.Vital signs (HR, BP, SpO2) were recorded at the beginning and at the end of each session, as well as monitored before, during and after the elliptical exercise. During the training, the vital signs were recorded on the first 30 seconds of each resting interval.
* The aerobic associate resisted physical training consisted of thirty minutes oa aerobic training at 60-70% of work rate obtained in CPT and subsequently three sets of fifteen repetitions of resistance training in lower limbs on leg press with an intensity of 40-60% of one repetition maximum test.

ELIGIBILITY:
Inclusion Criteria:

* Experimental Group:

  * Patients with clinical and spyrometric diagnosis of COPD presenting FEV1/FVC < 70% and FEV1 < 80% predicted by pulmonary function observed and were classified as patients with moderate to very severe obstruction (GOLD, 2010).
  * Clinically stable with no history infection or exacerbation of the respiratory symptoms or change in medication for two months preceding the study.
  * Patients were non oxygen dependent, smokers or former smokers.
  * No subject in the COPD group had ever participated in a pulmonary rehabilitation program (i.e., sedentary during the year preceding admission to the study).
  * Adherence to the individually prescribed treatment regimen.
* Control Group:

  * Pulmonary Function normal.
  * Subjects in the control group were free of chronic pulmonary, cardiovascular, immune, and metabolic disease.
  * Healthy controls who were sedentary during the year preceding admission to the study.

Exclusion Criteria:

* Patients with clinical diagnosis of COPD presenting FEV1/FVC ≥ 70% FEV1 ≥ 80% predicted (GOLD, 2010).
* Malignancy, orthopedic or neurological conditions affecting the ability to exercise, peripheral arterial disease, clinically apparent heart failure, and/or any renal, hepatic or inflammatory disease.
* Changed the type of medication during the study.
* Uncontrolled hypertension patients.
* Peripheral oxygen saturation below 90% at rest.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-01; Primary Completion 2010-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Effect of aerobic and resisted physical training and interval physical training on oxygen uptake and heart rate on-kinetics in patients with COPD. | baseline and 6 weeks
  The kinetic analysis was measured before and after interval physical training and aerobic and resisted physical training by Cardiopulmonary Exercise Testing (CPT; Incremental symptom-limited exercise testing), Constant-load exercise test in cycle ergometer and Constant-load exercise test in elliptical equipament. The on-transient (first 180 seconds) response of VO2 and HR was modeled according to a monoexponencial fit.

SECONDARY OUTCOMES:
Change in oxygen consumption, minute ventilation, ventilatory limitation, pulmonary carbon dioxide output, metabolic rate. | baseline and 6 weeks
  It was evaluated through a MedGraphics VO2000 metabolic system which was operated via computer with Aerograph software and store the signals with the three breath method at the peak of CPT and in the peak of Constant-load exercise test in cycle ergometer and Constant-load exercise test in elliptical equipament before and after interval physical training and aerobic and resisted physical training
Change in oxygenation | baseline and 6 weeks
  It was evaluated through a Nonin® (modelo 2500, Minneapolis, Mn, USA)wrist pulse oxymeter at the peak of CPT and peak of Constant-load exercise test in cycle ergometer and Constant-load exercise test in elliptical before and after aerobic/resisted physical training and interval physical training in elliptical equipament.
Change in heart rate and heart rate reserve | baseline and 6 weeks
  It was evaluated through a Polar® cardiofrequency (Polar® FS2cTM Kempele, Finland) at the peak of CPT and peak of Constant-load exercise test in cycle ergometer and Constant-load exercise test in elliptical before and after aerobic/resisted physical training and interval physical training in elliptical equipament.
Change in dyspnea and perceived discomfort in lower limbs | baseline and 6 weeks
  It was evaluated through a Borg scale (BORG, 1982) at the peak of CPT and peak of Constant-load exercise test in cycle ergometer and Constant-load exercise test in elliptical before and after aerobic/resisted physical training and interval physical training in elliptical equipament.
Change in quality of life and Daily Life Activities | baseline and 6 weeks
  It was evaluated through a St George's Respiratory Questionnaire (SGRQ) and London Chest Activity of Daily Living Scale (LCADL)(PITTA et al, 2008; CARPES et al, 2008) before and after aerobic/resisted physical training and interval physical training in elliptical equipament.
Change in Body composition | baseline and 6 weeks
  It was evaluated through a body composition monitor, evaluated weight, body fat percentage, muscle mass free, basal metabolic rate, bone mass and total body water percentage before and after aerobic/resisted physical training and interval physical training in elliptical equipament.
Change in BODE Index | baseline and 6 weeks
  It was evaluated through multidimensional index comprising of Body Mass Index (BMI), degree of airway obstruction (FEV1), functional dyspnea (MRC dyspnea scale), and exercise capacity by the 6 minute walk test (6MWT). For calculation of the BODE index, we used an empirical model as previously described by Celli et al. (2004), before and after aerobic/ resisted physical training and interval physical training in elliptical equipament.
Change in exercise capacity | baseline and 6 weeks
  It was evaluated through of performance obtained at the peak of CPT and in the peak of Constant-load exercise test in cycle ergometer and Constant-load exercise test in elliptical equipament before and after interval physical training and aerobic and resisted physical training

CONTACTS AND LOCATIONS:
Overall Officials: Bruna V Pessoa, Ms, Principal Investigator — Universidade Federal de Sao Carlos
Locations (1):
- Federal University of sao Carlos, São Carlos, São Paulo, Brazil

REFERENCES:
- [Result] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Result] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893
- [Result] Dourado VZ, Tanni SE, Vale SA, Faganello MM, Sanchez FF, Godoy I. Systemic manifestations in chronic obstructive pulmonary disease. J Bras Pneumol. 2006 Mar-Apr;32(2):161-71. doi: 10.1590/s1806-37132006000200012. English, Portuguese. PMID 17273586
- [Result] Rabe KF, Hurd S, Anzueto A, Barnes PJ, Buist SA, Calverley P, Fukuchi Y, Jenkins C, Rodriguez-Roisin R, van Weel C, Zielinski J; Global Initiative for Chronic Obstructive Lung Disease. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease: GOLD executive summary. Am J Respir Crit Care Med. 2007 Sep 15;176(6):532-55. doi: 10.1164/rccm.200703-456SO. Epub 2007 May 16. PMID 17507545
- [Result] Knudson RJ, Lebowitz MD, Holberg CJ, Burrows B. Changes in the normal maximal expiratory flow-volume curve with growth and aging. Am Rev Respir Dis. 1983 Jun;127(6):725-34. doi: 10.1164/arrd.1983.127.6.725. PMID 6859656
- [Result] Casaburi R, Porszasz J, Burns MR, Carithers ER, Chang RS, Cooper CB. Physiologic benefits of exercise training in rehabilitation of patients with severe chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 1997 May;155(5):1541-51. doi: 10.1164/ajrccm.155.5.9154855.
- [Result] Nasis IG, Vogiatzis I, Stratakos G, Athanasopoulos D, Koutsoukou A, Daskalakis A, Spetsioti S, Evangelodimou A, Roussos C, Zakynthinos S. Effects of interval-load versus constant-load training on the BODE index in COPD patients. Respir Med. 2009 Sep;103(9):1392-8. doi: 10.1016/j.rmed.2009.03.003. Epub 2009 Apr 5. PMID 19349153
- [Result] Vogiatzis I, Nanas S, Roussos C. Interval training as an alternative modality to continuous exercise in patients with COPD. Eur Respir J. 2002 Jul;20(1):12-9. doi: 10.1183/09031936.02.01152001. PMID 12166558
- [Result] Kortianou EA, Nasis IG, Spetsioti ST, Daskalakis AM, Vogiatzis I. Effectiveness of Interval Exercise Training in Patients with COPD. Cardiopulm Phys Ther J. 2010 Sep;21(3):12-9. PMID 20957074
- [Result] Franssen FM, Broekhuizen R, Janssen PP, Wouters EF, Schols AM. Effects of whole-body exercise training on body composition and functional capacity in normal-weight patients with COPD. Chest. 2004 Jun;125(6):2021-8. doi: 10.1378/chest.125.6.2021. PMID 15189917
- [Result] Spruit MA, Gosselink R, Troosters T, De Paepe K, Decramer M. Resistance versus endurance training in patients with COPD and peripheral muscle weakness. Eur Respir J. 2002 Jun;19(6):1072-8. doi: 10.1183/09031936.02.00287102. PMID 12108859
- [Result] Panton LB, Golden J, Broeder CE, Browder KD, Cestaro-Seifer DJ, Seifer FD. The effects of resistance training on functional outcomes in patients with chronic obstructive pulmonary disease. Eur J Appl Physiol. 2004 Apr;91(4):443-9. doi: 10.1007/s00421-003-1008-y. Epub 2003 Nov 25. PMID 14639479
- [Result] Misic MM, Valentine RJ, Rosengren KS, Woods JA, Evans EM. Impact of training modality on strength and physical function in older adults. Gerontology. 2009;55(4):411-6. doi: 10.1159/000227804. Epub 2009 Jul 3. PMID 19590159
- [Result] Egana M, Donne B. Physiological changes following a 12 week gym based stair-climbing, elliptical trainer and treadmill running program in females. J Sports Med Phys Fitness. 2004 Jun;44(2):141-6. PMID 15470311
- [Result] Kim JK, Nho H, H Whaley M. Inter-modal comparisons of acute energy expenditure during perceptually based exercise in obese adults. J Nutr Sci Vitaminol (Tokyo). 2008 Feb;54(1):39-45. doi: 10.3177/jnsv.54.39. PMID 18388406
- [Result] Burnfield JM, Shu Y, Buster T, Taylor A. Similarity of joint kinematics and muscle demands between elliptical training and walking: implications for practice. Phys Ther. 2010 Feb;90(2):289-305. doi: 10.2522/ptj.20090033. Epub 2009 Dec 18. PMID 20022994
- [Result] Lu TW, Chien HL, Chen HL. Joint loading in the lower extremities during elliptical exercise. Med Sci Sports Exerc. 2007 Sep;39(9):1651-8. doi: 10.1249/mss.0b013e3180dc9970. PMID 17805099
- [Result] Puente-Maestu L, Sanz ML, Sanz P, Nunez A, Gonzalez F, Whipp BJ. Reproducibility of the parameters of the on-transient cardiopulmonary responses during moderate exercise in patients with chronic obstructive pulmonary disease. Eur J Appl Physiol. 2001 Sep;85(5):434-41. doi: 10.1007/s004210100486. PMID 11606012
- [Result] Chiappa GR, Borghi-Silva A, Ferreira LF, Carrascosa C, Oliveira CC, Maia J, Gimenes AC, Queiroga F Jr, Berton D, Ferreira EM, Nery LE, Neder JA. Kinetics of muscle deoxygenation are accelerated at the onset of heavy-intensity exercise in patients with COPD: relationship to central cardiovascular dynamics. J Appl Physiol (1985). 2008 May;104(5):1341-50. doi: 10.1152/japplphysiol.01364.2007. Epub 2008 Mar 20. PMID 18356477
- [Result] Laveneziana P, Valli G, Onorati P, Paoletti P, Ferrazza AM, Palange P. Effect of heliox on heart rate kinetics and dynamic hyperinflation during high-intensity exercise in COPD. Eur J Appl Physiol. 2011 Feb;111(2):225-34. doi: 10.1007/s00421-010-1643-z. Epub 2010 Sep 18. PMID 20852881
- [Result] Somfay A, Porszasz J, Lee SM, Casaburi R. Effect of hyperoxia on gas exchange and lactate kinetics following exercise onset in nonhypoxemic COPD patients. Chest. 2002 Feb;121(2):393-400. doi: 10.1378/chest.121.2.393. PMID 11834648
- [Result] Chiappa GR, Queiroga F Jr, Meda E, Ferreira LF, Diefenthaeler F, Nunes M, Vaz MA, Machado MC, Nery LE, Neder JA. Heliox improves oxygen delivery and utilization during dynamic exercise in patients with chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2009 Jun 1;179(11):1004-10. doi: 10.1164/rccm.200811-1793OC. Epub 2009 Mar 19. PMID 19299497
- [Result] Poole DC, Ferreira LF, Behnke BJ, Barstow TJ, Jones AM. The final frontier: oxygen flux into muscle at exercise onset. Exerc Sport Sci Rev. 2007 Oct;35(4):166-73. doi: 10.1097/jes.0b013e318156e4ac. PMID 17921784
- [Result] Cerretelli P, Shindell D, Pendergast DP, Di Prampero PE, Rennie DW. Oxygen uptake transients at the onset and offset of arm and leg work. Respir Physiol. 1977 Jun;30(1-2):81-97. doi: 10.1016/0034-5687(77)90023-8. PMID 877453
- [Result] Williamson JW, Raven PB, Whipp BJ. Unaltered oxygen uptake kinetics at exercise onset with lower-body positive pressure in humans. Exp Physiol. 1996 Jul;81(4):695-705. doi: 10.1113/expphysiol.1996.sp003970. PMID 8853277
- [Result] Hughson RL, Cochrane JE, Butler GC. Faster O2 uptake kinetics at onset of supine exercise with than without lower body negative pressure. J Appl Physiol (1985). 1993 Nov;75(5):1962-7. doi: 10.1152/jappl.1993.75.5.1962. PMID 8307846
- [Result] Egana M, O'Riordan D, Warmington SA. Exercise performance and VO2 kinetics during upright and recumbent high-intensity cycling exercise. Eur J Appl Physiol. 2010 Sep;110(1):39-47. doi: 10.1007/s00421-010-1466-y. Epub 2010 Apr 13. PMID 20386919
- [Result] Koga S, Shiojiri T, Shibasaki M, Kondo N, Fukuba Y, Barstow TJ. Kinetics of oxygen uptake during supine and upright heavy exercise. J Appl Physiol (1985). 1999 Jul;87(1):253-60. doi: 10.1152/jappl.1999.87.1.253. PMID 10409583
- [Result] Leyk D, Essfeld D, Hoffmann U, Wunderlich HG, Baum K, Stegemann J. Postural effect on cardiac output, oxygen uptake and lactate during cycle exercise of varying intensity. Eur J Appl Physiol Occup Physiol. 1994;68(1):30-5. doi: 10.1007/BF00599238. PMID 8162920
- [Result] Rossiter HB, Ward SA, Kowalchuk JM, Howe FA, Griffiths JR, Whipp BJ. Effects of prior exercise on oxygen uptake and phosphocreatine kinetics during high-intensity knee-extension exercise in humans. J Physiol. 2001 Nov 15;537(Pt 1):291-303. doi: 10.1111/j.1469-7793.2001.0291k.x. PMID 11711581
- [Result] Schneider DA, Wing AN, Morris NR. Oxygen uptake and heart rate kinetics during heavy exercise: a comparison between arm cranking and leg cycling. Eur J Appl Physiol. 2002 Nov;88(1-2):100-6. doi: 10.1007/s00421-002-0690-5. Epub 2002 Sep 18. PMID 12436276
- [Result] Fukuoka Y, Endo M, Kagawa H, Itoh M, Nakanishi R. Kinetics and steady-state of VO2 responses to arm exercise in trained spinal cord injury humans. Spinal Cord. 2002 Dec;40(12):631-8. doi: 10.1038/sj.sc.3101383. PMID 12483496
- [Result] Crouter SE, Antczak A, Hudak JR, DellaValle DM, Haas JD. Accuracy and reliability of the ParvoMedics TrueOne 2400 and MedGraphics VO2000 metabolic systems. Eur J Appl Physiol. 2006 Sep;98(2):139-51. doi: 10.1007/s00421-006-0255-0. Epub 2006 Aug 3. PMID 16896734
- [Result] Bell C, Paterson DH, Kowalchuk JM, Padilla J, Cunningham DA. A comparison of modelling techniques used to characterise oxygen uptake kinetics during the on-transient of exercise. Exp Physiol. 2001 Sep;86(5):667-76. doi: 10.1113/eph8602150. PMID 11571496
- [Result] Engelen M, Porszasz J, Riley M, Wasserman K, Maehara K, Barstow TJ. Effects of hypoxic hypoxia on O2 uptake and heart rate kinetics during heavy exercise. J Appl Physiol (1985). 1996 Dec;81(6):2500-8. doi: 10.1152/jappl.1996.81.6.2500. PMID 9018498
- [Result] Berger NJ, Tolfrey K, Williams AG, Jones AM. Influence of continuous and interval training on oxygen uptake on-kinetics. Med Sci Sports Exerc. 2006 Mar;38(3):504-12. doi: 10.1249/01.mss.0000191418.37709.81. PMID 16540838
- [Result] Puente-Maestu L, Tena T, Trascasa C, Perez-Parra J, Godoy R, Garcia MJ, Stringer WW. Training improves muscle oxidative capacity and oxygenation recovery kinetics in patients with chronic obstructive pulmonary disease. Eur J Appl Physiol. 2003 Feb;88(6):580-7. doi: 10.1007/s00421-002-0743-9. Epub 2002 Nov 30. PMID 12560958